CLINICAL TRIAL: NCT00140335
Title: Evaluation of a Handwashing Promotion Program in Chinese Elementary Schools
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: Procter and Gamble (Industry); Centers for Disease Control and Prevention, China (Other Government); Fujian Province CDC (Unknown)
Responsible Party: Anna Bowen, CDC
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CDC-NCID-4427
Record Dates: First submitted 2005-08-30; First posted 2005-09-01 (Estimated); Last update posted 2010-03-09 (Estimated); Status verified 2010-03

CONDITIONS: Communicable Diseases
Keywords: handwashing; communicable diseases; health education
MeSH Terms: conditions — Communicable Diseases; Health Education | interventions — Hand Disinfection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: handwashing

SUMMARY:
The purpose of this study is to determine the effects of a commercial hand washing promotion program on hygiene knowledge, attitudes, and practices, and on health outcomes such as reported infectious illnesses and school absences.

DETAILED DESCRIPTION:
Diarrheal and respiratory diseases cause 3.8 million deaths annually among children in the developing world. Reduced rates of these diseases have been measured during intensive, home-based handwashing interventions. We evaluated a school-based handwashing program for 1st grade students to determine whether a more scalable intervention could also reduce illness rates, and impact hygiene knowledge and attitudes.

Thirty schools from each of 3 counties in Fujian Province, China, were randomized to one of the following groups: a) control; b) standard intervention, which included a handwashing program (1 hour of hygiene instruction and 1 soap sample kit per pupil); or c) expanded intervention, which included the handwashing program, soap for school sinks and 1 peer hygiene monitor per class. Teachers collected illness symptom information from students weekly and recorded student absences daily between January and April, 2005. Mean illness and absence rates were calculated for each school. Students were given a knowledge, attitudes, and practices questionnaire before the intervention and again 5 months later.

ELIGIBILITY:
Inclusion Criteria:

* school has running water

Exclusion Criteria:

* school has not previously received commercial handwashing promotion program

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 5000
Dates: Start 2004-12; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
student illness rates
student absence rates

SECONDARY OUTCOMES:
teacher illness rate
changes in student hygiene knowledge
changes in student hygiene attitudes
changes in school water use

CONTACTS AND LOCATIONS:
Overall Officials: Anna B Bowen, MD, MPH, Study Director — Centers for Disease Control and Prevention
Locations (1):
- Fujian Province CDC, Fuzhou, Fujian, China